



# Study Protocol

Study Title: Choice of Inhalation Device in Asthma and COPD

**Study Acronym:** CIDAC **Phase of Development:** NA

**Protocol Number:** 

Protocol Version and Date: Version number 1, 05/03/2021

EudraCT Registry Number: (ter info: zal gebeuren via studieloket UZ Brussel zodra ik

goedkeuring ethisch committee heb)

ClinicTrials.gov Registry Number: (idem zie boven)

**Indication:** obstructive lung disease

Investigational product or Medical Device: NA

**Sponsor: NA** 

Coordinating/Principal Investigator: Laure Vandermeersch

The information contained in this document is the property of the Sponsor/Coordinating Investigator and may not be reproduced, published or disclosed to others without written authorization of the Sponsor/Coordinating Investigator.

### PROTOCOL SIGNATURE PAGE

Protocol Version and date: Version number 1, 5 March 2021

Protocol Title: Choice of inhalation device in asthma and COPD patients

**Sponsor:** This study is an academic study and has no sponsor.

**Principal Investigator:** Laure Vandermeersch

#### I agree:

- to assume responsibility for the proper conduct of this study
- to conduct the study in compliance with this protocol and any future amendments
- not to implement any deviations from or changes to the protocol without prior review and written approval from the Ethics Committee, except where necessary to eliminate an immediate hazard to the subjects, or for administrative aspects of the study (where permitted by all applicable regulatory requirements)
- that I am thoroughly familiar with the appropriate use of the investigational drug, as described in this protocol
- to ensure that all persons assisting me with the study are adequately informed about the investigational drug and their study-related duties and functions as described in the protocol
- that I am aware of and will comply with the current good clinical practice (GCP) guidelines and ethical principles outlined in the Declaration of Helsinki
- to conduct the study in accordance with all applicable laws and regulations

| Printed name | Signature | Date |
|--------------|-----------|-------|
| Printed name | Signature | 17816 |





## **Table of Contents**

| 1 | Tria | Trial Registration/Protocol Summary6 | |
|---|---|---|---|
| 2 | Prot | Protocol Version History | |
| 3 | Spoi | Sponsor/Coordinating Investigator Information | |
| 4 | List | of Abbreviations | 8 |
| 5 Introduction | | | 8 |
| | 5.1 | Overview of Disease Pathogenesis | 8 |
| | 5.2 | Epidemiology | 9 |
| | 5.3 | Current Treatments | 9 |
| | 5.4 | Study Rationale and Purpose | 10 |
| | 5.5 | Rationale for Study Design | 11 |
| | 5.6 | Rationale for Dose and Regimen/Schedule Selection | 11 |
| 6 | Stud | dy Schematic and Schedule of Activities | 12 |
| | 6.1 | Study Schematic | 12 |
| | 6.2 | Study Activities | 12 |
| 7 | Stud | dy Objectives and Endpoints | 13 |
| | 7.1 | Primary Objective | 13 |
| | 7.2 | Secondary Objectives | 13 |
| | 7.3 | Endpoints | 14 |
| 8 | Inve | stigational Plan | 14 |
| | 8.1 | Overall Study Design | 14 |
| | 8.2<br>8.2.1<br>8.2.2<br>8.2.3<br>8.2.4<br>8.2.5 | Treatment Period | 14<br>14<br>14 |
| 9 | Sele | ction of Subjects | 14 |
| | 9.1 | Selection of Study Population | 14 |
| | 9.2 | Inclusion Criteria | 14 |
| | 9.3 | Exclusion Criteria | 14 |





| | 9.4 | Contraception/Pregnancy Avoidance | 15 |
|---|---|---|---|
| 10 | ) Scre | ening and Randomization | 15 |
| | 10.1 | Screening and Enrollment | 15 |
| | 10.2 | Randomization | 15 |
| | 10.3 | Blinding Procedures | 15 |
| 11 | Inter | ventions/Treatment | 16 |
| | 11.1 | Treatments Administered | |
| | 11.2 | Product Characteristics | |
| | 11.3 | Randomization and Stratification | |
| | 11.4 | Direction of Administration | 16 |
| | 11.5 | Dosing Regimen | 16 |
| | 11.5 | 1 Dose Modifications and Dose Delay | 16 |
| | 11.5 | 2 Treatment Interruption and Treatment Discontinuation | 16 |
| | 11.6 | Treatment Compliance | 16 |
| | 11.7 | Study Drug or Medical Device Accountability | 16 |
| | 11.8 | Storage, Packaging and Labeling | 16 |
| | 11.9 | Blinding | 16 |
| | 11.10 | Prior and Concomitant Medication | 16 |
| | 11.11 | Non-Drug Therapies | 16 |
| | 11.12 | Prohibited Medication | |
| | 11.13 | Prohibited Procedures | 16 |
| | 11.14 | Other Interactions | 16 |
| | 11.15 | Study Disposal and Destruction | 16 |
| | 11.16 | Known Undesirable Effects of Study Drug | 16 |
| 12 | 2 Stud | y Assessments and Procedures | . 16 |
| | 12.1 | Study Assessments | 17 |
| | 12.1 | | |
| | 12.1 | | |
| | 12.1 | 3 Run-In | 17 |
| | 12.1. | | |
| | 12.1. | · | |
| | 12.1. | , and the state of | |
| | 12.1. | | |
| | 12.1.<br>12.1. | · | |
| | 14.1. | O OHOOHEGUIEU VIOIG | 17 |





| | 12.2 | | essment Types | |
|---|---|---|---|---|
| | 12.2 | | Efficacy Assessment | |
| | 12.2 | | Safety and Tolerability Assessments | |
| | 12.2 | | Physical Examination | |
| | 12.2<br>12.2 | | Vital Signs, Height, Weight | |
| | 12.2 | | ECG | |
| | 12.2 | .0 | Laboratory Evaluation | 10 |
| 13 | Safe | ty Mc | nitoring and Reporting1 | 8 |
| | 13.1 | | erse Events | |
| | 13.1 | | Definitions and Reporting | |
| | 13.1 | | Reporting Period | |
| | 13.1 | .3 | Laboratories Test Abnormalities | 18 |
| | 13.2 | Serio | ous Adverse Events | 18 |
| | 13.2 | | Definitions | |
| | 13.2 | | Immediate Reporting | |
| | 40.0 | _ | | |
| | 13.3 | | pected Unexpected Serious Adverse Events (SUSAR) | |
| | 13.3<br>13.3 | | Definitions | |
| | 13.3 | .∠ | Reporting | 19 |
| | 13.4 | Othe | r safety data requiring an immediate declaration | 19 |
| | 13.5 | | edures for Handling Special Situations | |
| | 13.5 | | Pregnancy | |
| | 13.5 | .2 | Overdose Management | 19 |
| | 13.6 | Δnnı | ual Safety Report | 10 |
| | 10.0 | Allite | di Galoty Noport | , , |
| 14 | Data | a Coll | ection and Management 1 | 9 |
| | 14.1 | | toring | 19 |
| | 14.1 | | Composition of data monitoring committee | |
| | 14.1 | .2 | Interim analysis | 19 |
| | 14.2 | Data | Collection | 19 |
| | 14.3 | Data | base Management and Quality Control | 19 |
| | 14.4 | Stati | stical Considerations and Data Analysis | 10 |
| | 14.4 | Stati | Silcal Considerations and Data Analysis | 13 |
| 15 | Ethi | cal Co | onsiderations2 | 20 |
| | 15.1 | | al conduct of the study | |
| | 15.1 | | Declaration of Helsinki | |
| | 15.1 | .2 | Ethics Committee | 20 |
| | 15.2 | Infor | med Consent | 20 |
| | 70.2 | 1111011 | 100 0010011 | -0 |
| | 15.3 | Patie | ent and Study Data Protection | 20 |
| | 45 4 | | | ~ ~ |
| | 15.4 | Subj | ect Identification | 20 |
| 16 | Fina | nce a | nd Insurance | )<br>() |
| | iiia | cc a | | |
| 17 | Repo | orting | gand Dissemination | <u>'</u> 1 |





| 18 | Conflict of Interest Statement | 21 |
|----|--------------------------------|------|
| 19 | Tables and Figures | . 22 |
| 20 | References | 73 |





## 1 Trial Registration/Protocol Summary

| Information | |
|---|---|
| EudraCT number: | Application for registration in a clinical trial registry will be done after obtaining |
| Date of registration: | approval from the ethics committee |
| ClinicalTrials.gov: | Please see previous line |
| Official Title: | Choice of inhalation device in asthma and COPD |
| Study Phase/Type: | Single center, single visit cross-sectional interventional study without device or investigational product. |
| Condition: | Asthma and COPD (Chronic Obstructive Pulmonary Disease) |
| Objectives: | To identify patient/inhalation device mismatch by using objective measurements. |
| Investigational Product or Medical Device: | NA NA |
| Interventions: | The intervention will be a three-step evaluation. Patients will perform a deep voluntary inspiration. This inspiration will be assessed by the investigator. Secondly, the peak inspiratory flow will be measured over 5 different resistances with an In-check Dial device. Subsequently, patients will receive education about good coordination technique, which is necessary for the optimal use of pressured metered dose inhalers (pMDIs). By using a placebo pMDI, the investigator will assess the coordination of the patient. The evaluation of voluntary deep inspiration, PIF's and coordination will be by pass or fail evaluation. |
| Endpoints: | To assess if the choice of inhaler device category differs when based on objective assessments, as compared to the choice made by the treating physician (during routine clinical practice), which is primarily based on subjective evaluation. |
| Study population: | Asthma and COPD patients treated with inhaled medications. Subjects will be recruited in the respiratory outpatient clinic in UZ Brussel after a scheduled consultation with their pulmonologist. |
| Number of patients: | 40 COPD patients (GOLD II-IV); 20 patients with severe asthma, 40 patients with asthma aged ≥ 70y, 40 patients with mild-to moderate asthma aged < 70y |
| Overview of | Single center, single visit cross-sectional interventional study without device or |
| study design: | investigational product |
| Statistical | Descriptive analysis will be used to describe the prevalence patient/device |
| Considerations: | mismatch. Multiple regression analysis will be performed to identify patient characteristics associated with inability to use the 3 main classes of inhalation devices respectively. Due to the exploratory nature of this study, no formal power calculation can be performed. |
| Sponsor: | This study is an academic study and has no sponsor. |
| Inclusion Criteria: | <ul> <li>COPD patients (GOLD II-IV)</li> <li>Patients with severe asthma</li> <li>Patients with asthma aged ≥ 70y</li> <li>Patients with mild-to moderate asthma aged &lt; 70y</li> </ul> |
| Exclusion Criteria: | <ul> <li>Patients with asthma or COPD not on inhaled therapy for maintenance treatment</li> <li>Patients younger than 18y</li> <li>Patients unable to give their informed consent due to mental or physical disability</li> <li>Patients who don't speak Dutch or French</li> </ul> |
| Target Date of first | To be determined. Probably Q4 2021. |
| enrolment: | |





Target sample size: No target sample size calculation could be performed due to exploratory nature of the study (please see above)





## 2 Protocol Version History

| Version No. | Release Date | Summary of Changes |
|-------------|--------------|--------------------|

## 3 Sponsor/Coordinating Investigator Information

Coordinating Investigator (promotor): Prof. Dr. Eef Vanderhelst

Sponsor: NA

Principal Investigator Laure Vandermeersch

Co-investigators: Prof. Dr. Eef Vanderhelst, Dr. Shane Hanon (co-promotor), Mr Daniël

Schuermans, Mss Cindy Zienebergh Additional co-researchers: NA

Statistician

Laboratory (ies): NA Pharmacy: NA

Study Coordinator; Daniël Schuermans

Study sites and co-investigators; respiratory outpatient clinic UZ Brussel

### 4 List of Abbreviations

COPD = Chronic Obstructive Pulmonary Disease
FEV1 = Forced Expiratory Volume in one second
FVC = Forced Vital Capacity
ICS = Inhaled corticosteroids
LABA = long acting beta-agonists
LAMA = long acting muscarinic antagonists
GOLD = Global Initiative for Chronic Obstructive Lung Disease
GINA = Global Initiative for Asthma

GINA = GIODAI IIIILIALIVE IOI ASLIIIII

## 5 Introduction

### 5.1 Overview of Disease Pathogenesis

### Pathogenesis of asthma

Asthma is a heterogeneous disease, which is normally characterized by the presence of chronic airway inflammation. Asthma is defined by the history of respiratory symptoms such as shortness of breath, wheeze, cough, chest tightness. These symptoms can fluctuate over time and in intensity in combination with a variable expiratory airflow limitation. (1)

### Pathogenesis of COPD

Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases





an influenced by host factors including abnormal lung development. Significant comorbidities may have an impact on morbidity and mortality.

The most common respiratory symptoms of COPD are cough and/or sputum production, dyspnea. Underreporting of these symptoms by patients can occur.

The most important risk factor for COPD is tobacco smoking. Other environmental exposures such as air pollution and biomass fuel exposure may contribute. (2)

### 5.2 Epidemiology

### Epidemiology of asthma

Currently, 4.3% of the population worldwide has asthma. The prevalence of asthma in the United States is 8.4%. The prevalence of asthma is on the rise. Asthma is more prevalent in black than in white persons. It is remarkable that the prevalence of asthma decreases with each successive higher poverty level group. Asthma has a significant impact on morbidity and mortality. (3)

### **Epidemiology of COPD**

The global prevalence of physiologically defined chronic obstructive pulmonary disease (COPD) in adults aged >40 years is approximately 9-10 per cent. (4)

The worldwide prevalence of chronic obstructive pulmonary disease (COPD) in adults older than 40 years old is approximately 9-10%. COPD is the fifth leading cause of years lost through early mortality or handicap (disability-adjusted life years). Country, sex and age are factors that influence the prevalence of COPD. (2)

#### 5.3 Current Treatments

#### Treatment of asthma

The current pharmacological treatment of asthma consists of the stepwise approach by GINA. The goal is to optimize the personalized asthma management by assessing, adjusting and reviewing the response to treatment.

The treatment depends on the number of step of GINA. The 5 different GINA steps are characterized by different treatments. Inhaled corticosteroids (ICS), short acting  $\beta$ 2- agonists (SABA) and long acting  $\beta$ 2 agonists (LABA)

There are 3 different types of inhalers: dry powder inhalers (DPI), pressurized metered dose inhaler (pMDI) and soft mist inhalers (SMI).

SMI's and pMDI's can be used in combination with an inhalation chamber. (5)







Figure 1: treatment of asthma

#### Treatment of COPD

The treatment of COPD depends on the group guided by GOLD: group A, B, C or D. The corner stone of the pharmacological treatment consists of bronchodilatation: LABA (long acting beta-agonists), LAMA (long acting muscarinic antagonists). A triple therapy: ICS, LABA and LAMA, is recommended in COPD GOLD D patients. (6)

### 5.4 Study Rationale and Purpose

Inhalation therapy is the cornerstone therapy in asthma and COPD patients. Unfortunately, many errors are associated with the use of inhalers, which leads to poor outcome for patients. Problems with the use of pressurized metered dose inhalers were described shortly after the launch of pMDI and still persist today. The use of dry powder inhalers (DPI's) is also frequently associated with errors.

The most common errors in the use of pMDI's are incorrect coordination, insufficient depth and/or speed of inspiration and no postinhalation breath-hold in.

The post frequent DPI errors are no complete expiration before inhalation, incorrect preparation and lack of postinhalation breath-hold in.

The overall prevalence of poor technique was 31%, of acceptable technique 41% and of correct technique only 31%. It can be concluded that incorrect inhaler technique in asthma and COPD patients is unacceptably frequent. Over the past 40 years, the prevalence of correct inhaler technique has not improved. The lack of correct inhalation technique may be a major obstacle, which withholds patients from achieving optimal asthma or COPD control. (7)

Incorrect use of inhalers is associated with reduced disease control. The strongest associations have been found between incorrect inhaler technique and older age, lower schooling and lack of





instruction about the correct inhaler technique by healthcare workers. These associations are independently of the inhaler type. Poor inhaler use is most common in older ages, but can occur at all ages. The misuse of inhalers is associated with an elevated risk of hospitalization, visits to the emergency department, treatments with oral corticosteroids and antimicrobials, and poor disease control. Instruction by healthcare workers about the correct use of inhalers is the only modifiable factor that can be useful to reduce the prevalence of inhaler misuse. (8)

The choice of inhalation device is an important decision and is often as important as the medication put in the device to achieve optimal outcomes for patients with asthma or COPD. The optimization of treatment could be established by switching between devices instead of increasing or changing the pharmacological therapy. There are multiple differences between the various devices such as particle size, release mechanism, drug deposition and required inspiratory flow. Switching devices should never be done without the patient consent. A patient should feel comfortable with their device in order to use it properly, which makes that switching of device is a careful process in which the patient has to be involved. (9)

In conclusion, the purpose of the study is to identify patient/inhalation mismatch by using objective measurements.

### 5.5 Rationale for Study Design

All assessments can be made on the spot following the consultation, which allows a cross sectional design.

5.6 Rationale for Dose and Regimen/Schedule Selection NA





## 6 Study Schematic and Schedule of Activities

### 6.1 Study Schematic

| <b>Characteristics of the study</b> | |
|---|---|
| Informed consent procedure: Inclusion criteria: | <ul> <li>Available in Dutch and French</li> <li>Signature and date written by participant</li> <li>COPD patients (GOLD II-IV)</li> </ul> |
| | <ul> <li>Patients with severe asthma</li> <li>Patients with asthma aged ≥ 70y</li> <li>Patients with mild-to moderate asthma aged &lt; 70y</li> </ul> |
| Exclusion criteria: | <ul> <li>Patients with asthma or COPD not on inhaled therapy for maintenance treatment</li> <li>Patients younger than 18y</li> <li>Patients unable to give their informed consent due to mental or physical disability</li> <li>Patients who don't speak French or Dutch</li> </ul> |
| Collection of data form patient file: | <ul> <li>Choice of inhaler by physician (current inhaled maintenance treatment)</li> <li>GOLD grade and group (COPD patients)</li> <li>GINA treatment step (asthma patients)</li> <li>Smoking status</li> <li>Height</li> <li>Weight</li> <li>Age</li> <li>FEV<sub>1</sub>, FVC, PIF if available</li> <li>Oral corticosteroid maintenance dose</li> </ul> |
| Study assessments: | <ul> <li>Voluntary deep inhalation</li> <li>Peak inspiratory flows (PIF's)</li> <li>Coordination (through a placebo pMDI)</li> </ul> |
| Reporting to treating physician in case of patient/device mismatch | <ul> <li>To avoid prescription of inappropriate inhaler</li> </ul> |

### 6.2 Study Activities

The study will take place in the respiratory outpatient clinic. Patients will be invited to participate in the study after the consultation with the pulmonologist. All pulmonologists have a flowchart regarding the optimal choice of inhaler at their disposition.

Patients will be provided sufficient time to read the informed consent file and to ask questions about the study. After giving their informed consent they will be screened for eligibility by an





investigator. Demographic data and characteristics will be retrieved from the medical record (EMD) of study participants.

The intervention will consist of three different steps.

First, the patient will perform a deep voluntary inspiration. The patient's ability to perform this inspiration will be assessed and scored by the investigator.

Secondly, the peak inspiratory flows (PIF) will be measured with an In-check Dial device over 5 different resistances.

The minimal and optimal peak inspiratory flow rates (PIFRs) differ by device. A minimum flow of 30 L/min is required for most DPI's. The optimal flow varies from 30 L/min to 35, 45, 50, 60 or 65 L/min. (10)

Due to the fact that there is still discussion about the effectiveness of PIF's going from 30 to 60 L/min, an arbitrary cut-off value will be set at 45 L/min. This cut-off value for sufficient PIF will be measured over a moderate resistance to distinguish subtherapeutic from therapeutic levels. (11) If the patient reaches a PIF lower than 45 L/min, the patient will be asked to make a second attempt.

Subsequently, the patient will receive education about the correct coordination, which is necessary in the use of dose inhalers. The patient will be evaluated for sufficient actuation-inhalation coordination, through a placebo pMDI.

The evaluation of the voluntary deep inspiration, PIF and coordination will be by pass or fail evaluation. Subsequently, the fitness of a patient to use any of the three inhaler classes will be determined by using a diagram designed by a Belgian expert group (unpublished to date; courtesy of Didier Cataldo, ULiège).

If a mismatch between prescribed inhaler and suitable inhaler types is found, the treating physician of the patient will be informed. By doing so, we wish to avoid patients receiving prescriptions for inhalers that they cannot use properly.

## 7 Study Objectives and Endpoints

### 7.1 Primary Objective

To study the prevalence of patient/device mismatch based on objective assessments.

### 7.2 Secondary Objectives

To assess the proportion of patient/device mismatch per patient subgroup.

To assess the fail rates for each objective measurement separately for the entire study population and per patient group.

To correlate the fail rates for each objective measurement separately with patient's characteristics per patient subgroup and overall (age, sex, height, weight, FEV<sub>1</sub>, FVC, PIF, GOLD grade and group, smoking status, GINA treatment step, oral corticosteroid dose).





To correlate fail rates for each objective measurement with patient's characteristics.

7.3 Endpoints

Cfr 7.1 and 7.2

## 8 Investigational Plan

8.1 Overall Study Design

Cross sectional study design

- 8.2 Study Duration for Subjects
  - 8.2.1 Screening

Patients will be recruited following their consultation with their pulmonologist. The recruitment of the patients will take place in the respiratory outpatient clinic of UZ Brussel.

- 8.2.2 Treatment Period NA
- 8.2.3 Unscheduled Visit(s) NA
- 8.2.4 Early Study Termination NA
- 8.2.5 End of Study

The duration of the study for each individual patient will be around 5 to 10 minutes. Participation ends when the patient leaves the pulmonology division at the outpatient clinic.

## 9 Selection of Subjects

9.1 Selection of Study Population

The selection of study population will take place in the respiratory outpatient clinic in UZ Brussel. The patients will be recruited following their consultation with the pulmonologist.

- 9.2 Inclusion Criteria
- COPD patients (GOLD II-IV)
- Patients with severe asthma included in the Belgian Severe Asthma registry aged <70
- Patients with asthma of any severity aged  $\geq 70$ y
- Patients with mild-to moderate asthma aged < 70y
- 9.3 Exclusion Criteria
- Patients with asthma or COPD not on inhaled therapy for maintenance treatment
- Patients younger than 18y





- Patients unable to give their informed consent due to mental or physical disability
- Patients who don't speak French or Dutch
- 9.4 Contraception/Pregnancy Avoidance NA

## 10 Screening and Randomization

10.1 Screening and Enrollment

Patients who gave their informed consent will be screened for eligibility by an investigator.

- 10.2 Randomization NA
- 10.3 Blinding Procedures NA





## 11 Interventions/Treatment

### 11.1 Treatments Administered

The intervention consists of physiological measurements. No treatment, drug or product will be administered. No device will be tested. The In-check-dial-device and placebo pMDI are merely tools to perform the physiological measurements.

- 11.2 Product Characteristics NA
- 11.3 Randomization and Stratification NA
- 11.4 Direction of Administration NA
- 11.5 Dosing Regimen NA
  - 11.5.1 Dose Modifications and Dose Delay
  - 11.5.2 Treatment Interruption and Treatment Discontinuation
- 11.6 Treatment Compliance NA
- 11.7 Study Drug or Medical Device Accountability NA
- 11.8 Storage, Packaging and Labeling NA
- 11.9 Blinding NA
- 11.10 Prior and Concomitant Medication NA
- 11.11 Non-Drug Therapies NA
- 11.12 Prohibited Medication NA
- 11.13 Prohibited Procedures NA
- 11.14 Other Interactions NA
- 11.15 Study Disposal and Destruction NA
- 11.16 Known Undesirable Effects of Study Drug NA

## 12 Study Assessments and Procedures

Please see section 6.2: study activities





### 12.1 Study Assessments:

- 12.1.1 Screening cfr supra (6.2 and 10.1)
- 12.1.2 Baseline: NA
- 12.1.3 Run-In: NA
- 12.1.4 Treatment Period: NA
- 12.1.5 Follow-Up
- 12.1.6 End of Study

The study will end when the anticipated number of participants will be reached.

- 12.1.7 Re-screening NA
- 12.1.8 Early Termination NA
- 12.1.9 Unscheduled Visits NA

NA= not applicable for this cross-sectional study

### 12.2 Assessment Types

This study will assess physiological data (ability to perform a voluntary inhalation, PIF, and actuation-inhalation coordination with a pMDI). Cfr supra.





- 12.2.1 Efficacy Assessment NA
- 12.2.2 Safety and Tolerability Assessments NA
- 12.2.3 Physical Examination NA
- 12.2.4 Vital Signs, Height, Weight...

The height and weight of patients will be collected from the patient file.

- 12.2.5 ECG.... NA
- 12.2.6 Laboratory Evaluation NA
  - 12.2.6.1 Clinical Chemistry
  - 12.2.6.2 Hematology
  - 12.2.6.3 Urine Analysis
  - 12.2.6.4 Pharmacokinetics....

## 13 Safety Monitoring and Reporting

Patient safety during the assessments is monitored by the investigators. In the highly unlikely event of an adverse event (AE) or severe adverse event (SAE), this will be reported in the CRF and the treating physician will immediately be notified by the investigator.

The assessments of a deep inhalation, PIF maneuvers over a resistance and the use of a placebo pMDI do not differ from the maneuvers performed in daily life, when inhaler therapy is used by patients.

- 13.1 Adverse Events NA
  - 13.1.1 Definitions and Reporting

Reporting in the CRF

13.1.2 Reporting Period

Duration of the study for the individual patient

- 13.1.3 Laboratories Test Abnormalities: NA
- 13.2 Serious Adverse Events
  - 13.2.1 Definitions
  - 13.2.2 Immediate Reporting

Immediate reporting in the CRF and to the treating physician by the investigator





- 13.3 Suspected Unexpected Serious Adverse Events (SUSAR) NA
  - 13.3.1 Definitions
  - 13.3.2 Reporting
- 13.4 Other safety data requiring an immediate declaration NA
- 13.5 Procedures for Handling Special Situations NA
  - 13.5.1 Pregnancy
  - 13.5.2 Overdose Management
- 13.6 Annual Safety Report NA

### 14 Data Collection and Management

- 14.1 Monitoring
  - 14.1.1 Composition of data monitoring committee: NA
  - 14.1.2 Interim analysis: NA
- 14.2 Data Collection

By the investigator (from medical records and study assessments).

14.3 Database Management and Quality Control

The promotors and investigators from UZ Brussel's respiratory division assume database management and quality control.

### 14.4 Statistical Considerations and Data Analysis

The promotors and investigators from UZ Brussel's respiratory division will perform the statistical analysis, with the help of VUB statistician Professor Kurt Barbé.

The statistical plan was discussed during a meeting with professor Barbé (see below).

### Sample size calculation

This is a purely explorative study, since there is no a piori hypothesis to be confirmed. Hence, no formal sample size calculation is possible.

The findings of this study could later on be confirmed and assessed more extensively in larger dedicated studies.

For this study however, it is important that the patient groups be stratified according to their occurrence in society. We believe this will be the case when the in-and exclusion criteria for this study will be applied.





### Statistical analysis

Descriptive statistics will be used to describe the prevalence of patient/device mismatch for the entire study population.

The comparison of the prevalence of patient/device mismatch between patient subgroups and the comparison of the fail rates for each objective measurement separately between patient subgroups will be done by means of the Chi-square test and will be visualized in cross-tables.

To study correlations between patient characteristics (independent variables) and pass or fail rates for each of the three test criteria (dependent variables), box-plots will be used for continuous variables (for example weight and length), whereas the Chi-square test will be used for categorical variables (for example diagnosis, age expressed in years, GOLD stage and GOLD group).

### 15 Ethical Considerations

### 15.1 Ethical conduct of the study

### 15.1.1 Declaration of Helsinki

The study will be conducted in accordance with the principles and guidelines of the declaration of Helsinki.

### 15.1.2 Ethics Committee

Application for approval of this protocol by UZ Brussel's ethics committee is being prepared.

#### 15.2 Informed Consent

Patients will sign an informed consent before participating in the study. The informed consent will be available in Dutch and French.

### 15.3 Patient and Study Data Protection

This study will be performed in accordance with the standards applied by the UZ Brussel's Data Protection Officer.

Paper CRF's (source data) will be stored only in UZ Brussel's respiratory division. Anonymized data (excel file) will be stored on UZ Brussel's S-drive.

### 15.4 Subject Identification

Data will be anonymized before storage.

## 16 Finance and Insurance

The conduct of this academic study will be financed by UZ Brussel's respiratory division. An insurance will be taken out for this study.





## 17 Reporting and Dissemination

The principal investigator will report the results of the study in her master thesis. The results may also be presented at a scientific conference or be published. The investigators hold all publication rights.

## 18 Conflict of Interest Statement

The investigators have no conflicts of interest related to this study.





## 19 Tables and Figures



**Figure 1:** Diagram designed by a Belgian expert group: unpublished to date; used under permission of Prof. Dr. Didier Cataldo and courtesy of Prof. Dr. Didier Cataldo, University of Liège.

### Legend of the used colours in this diagram:

Green = optimal indication

Yellow = not indicated

Red = not indicated





### 20 References

- 1. Reddel Helen K et al. A summary of the new GINA strategy: a roadmap to asthma control. Eur Respir J. 2015; 46: 622-639
- 2. GOLD guidelines 2020, https://goldcopd.org/wp-content/uploads/2019/12/GOLD-2020-FINAL-ver1.2-03Dec19\_WMV.pdf
- 3. Loftus P, Wise S. Epidemiology of asthma. Curr Opin Otolaryngol Head Neck Surg. 2016 Jun; 24(3):245-9.
- 4. Vijayan V K. Chronic obstructive pulmonary disease. Indian J Med Res. 2013 Feb; 137 (2):251-69.
- 5. Gina Guidelines 2020, https://ginasthma.org/wp-content/uploads/2020/06/GINA-2020-report\_20\_06\_04-1-wms.pdf
- 6. Ferreira J et al. Optimal treatment sequence in COPD: Can a consensus be found? Revista Portuguesa de Pneumologia (English Edition). 2016 Jan-Feb; 22(1):39-49.
- 7. Sanchis J, Gich I, Pedersen S. Systematic Revies of Errors in Inhaler use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406.
- 8. Melani A et al. Inhaler mishandling remains common in real life and is associated with reduced disease control. Respir Med. 2011 Jun; 105(6):930-8.
- 9. Kaplan A, van Boven J. Switching Inhalers: A Practical Approach to keep on UR RADAR. Pulm. Ther. 2020 Dec;6(2):381-392.
- 10. Gosh S, Ohar J, Drummond M. Peak Inspiratory Flow Rate in Chronic Obstructive Pulmonary Disease: Implications for Dry Powder Inhalers. J Aerosol Med Pulm Drug Deliv. 2017 Dec 1; 30(6):381-387.
- 11. Janssens W et al. Inspiratory flow rate at different levels of resistance in elderly COPD patients. Eur Resp J 2008; 31:78-83.